CLINICAL TRIAL: NCT06492018
Title: Lay User Evaluation of the Panbio™ HCV Self Test in an EU Population
Status: Not yet recruiting | Type: Observational
Sponsor: Abbott Rapid Dx (Industry)
Responsible Party: Sponsor
Other Study IDs: SDRD-J-011-P
Record Dates: First submitted 2024-05-16; First posted 2024-07-09 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Hepatitis C
Keywords: Rapid diagnostic test; Antibodies to Hepatitis C Virus (HCV).; Self-test; Lay user
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Panbio™ HCV Self Test — Rapid diagnostic test (self-test and professional) plus laboratory reference tests
  Other Names: Fingerstick HIV testing (optional); Laboratory reference testing for HCV (immunoassays and PCR, CE marked)

SUMMARY:
This study is part of the performance evaluation to support the conformity assessment procedure for the use of fingerstick whole blood samples with Abbott's Panbio™ HCV Self Test device, as performed by lay users. The study will be conducted in accordance with the Commission Implementing Regulation (EU) 2022/1107 of 4 July 2022 laying down common specifications for certain class D in vitro diagnostic medical devices in accordance with Regulation (EU) 2017/746 of the European Parliament and of the Council and, to provide data to demonstrate the product is safe and effective for its intended use.

DETAILED DESCRIPTION:
Hepatitis C is a liver disease caused by the hepatitis C virus (HCV). The virus can cause both acute and chronic disease, ranging in severity from a mild illness lasting a few weeks to a serious, lifelong illness. Globally, around 50 million people per year are living with HCV, resulting in 244,000 deaths. The WHO estimates that only 36% of individuals chronically infected with HCV are diagnosed, and the WHO HCV targets include increasing the diagnoses to 90% by 2030. WHO guidelines, published in 2021, strongly recommend offering self-testing for HCV as an additional approach to HCV testing services.

The Panbio™ HCV Self Test, is a lateral flow test, designed for the qualitative detection of antibodies specific to HCV in finger-stick whole blood. The test is designed to be used by lay users and uses a sample volume of 10 µL. The professional use version test (Bioline™ HCV Test) is commercially available and has previously been clinically validated by the manufacturer, demonstrating a sensitivity of 99.3-100% and a specificity of 98.1-100%.

Evaluation of the test performance when used by professional users has been conducted, and evaluation of lay user sensitivity and specificity based on lay user populations outside the EU is being conducted. This study will demonstrate the test performance and usability of the test when used in a European lay user population. The study will be conducted at one recruiting hospital in Spain.

ELIGIBILITY:
Inclusion Criteria:

* Participant is aged 18 or over
* Participant agrees to all aspects of the study and is able and willing to provide informed consent / assent with parental consent.

Exclusion Criteria:

* Participant has already participated in this study on a previous occasion.
* Participant is deemed unfit for the study by the Investigator.
* Participant has a condition deemed unfit by the Investigator to safely perform or receive the test.
* Participant is a practising health-care professional or laboratory scientist / technician or has prior medical or laboratory training or experience
* Participant is currently enrolled in a study to evaluate an investigational drug or vaccine.
* Participant has a visual impairment that cannot be restored using glasses or contact lenses or is unable to read the Instructions for Use.
* Participant is unwilling or unable to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants with any known or suspected anti-HCV status may be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Lay user / professional user test result concordance | 5 months
  To assess the concordance between the Panbio™ HCV Self Test, as performed by lay users based on self-collected finger-stick samples, and the Panbio™ HCV Self Test performed by a trained health care worker, who also will collect the finger-stick sample required for the test and perform the test.
Lay user / laboratory test result concordance | 5 months
  To establish clinical performance (concordance with the reference test) for the Panbio™ HCV Self Test, as performed by lay users using finger-stick whole blood samples, when compared to reference testing using venous plasma samples.

SECONDARY OUTCOMES:
Labelling comprehension evaluation | 5 months
  To evaluate user experience and lay user participants' understanding of the test through a questionnaire. The participant questionnaire includes questions which are intended to evaluate the lay user's understanding of the Quick Reference Guide / Instructions for Use. Most questions have a Yes / No answer option, with free text possible. Some questions require a free text answer.
Results interpretation evaluation | 5 months
  To evaluate the lay users' understanding of static test results (mock devices).
Usability evaluation - lay user experience | 5 months
  To assess the usability of the Panbio™ HCV Self Test, as performed by lay users, based on a participant questionnaire evaluation by the lay user participant. The participant questionnaire includes questions to assess the lay users' experience when performing the test. Most questions have a Yes / No answer option, with free text possible. Some questions require a free text answer.
Usability evaluation - Self-test observer records | 5 months
  To assess the usability of the Panbio™ HCV Self Test, as performed by lay users based on a questionnaire evaluation by the study staff observer. In the observer questionnaire, particular attention will be paid to compliance regarding factors considered critical for the test, such as reading the IFU/ QRG and applying the correct test volume.
  The observer questionnaire is not reporting scores on a scale, but is recording observations regarding how the users complete each step. For each step, a question is asked whether the user conducted a certain procedure, and a Yes / No answer is requested, with Monitor Notes when applicable.
Lay user / professional user results interpretation concordance | 5 months
  To assess the concordance between the self-test results (obtained by the self-tester) when interpreted by the lay user and by the observer.

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Ryan, MD, PhD, Principal Investigator — Hospital Universitario Infanta Leonor
Locations (1):
- Hospital Universitario infanta Leonor, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No